CLINICAL TRIAL: NCT00047268
Title: Prospective Study of the Diagnosis and Treatment of Myelodysplastic Syndromes (MDS) in Childhood
Brief Title: Donor Stem Cell Transplant With or Without Chemotherapy in Treating Children With Primary Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Working Group of MDS in Childhood (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000257581; EWOG-MDS-98; EU-20218
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2007-07

CONDITIONS: Leukemia; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: juvenile myelomonocytic leukemia; childhood myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; chronic myelomonocytic leukemia
MeSH Terms: conditions — Leukemia; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Leukemia, Myelomonocytic, Chronic | interventions — Cytarabine; Mercaptopurine; Biopsy; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: cytarabine
Drug: mercaptopurine
Other: laboratory biomarker analysis
Procedure: allogeneic bone marrow transplantation
Procedure: biopsy
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor stem cell transplant helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. It is not yet known whether donor stem cell transplant is more effective with or without chemotherapy in treating primary myelodysplastic syndrome.

PURPOSE: This phase III trial is studying how well donor stem cell transplant given with chemotherapy works and compares it with donor stem cell transplant without chemotherapy in treating children with primary myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine, by a standard approach, the frequency of different FAB subtypes in children with primary myelodysplastic syndromes.
* Determine the frequency of cytogenetic and molecular abnormalities in these patients.
* Determine the survival of patients treated with allogeneic stem cell transplantation with or without induction chemotherapy.
* Determine the rate of complete remission in patients treated with these regimens.
* Determine the event-free survival of patients treated with these regimens.
* Determine the relapse rate, morbidity, and mortality of patients treated with these regimens.
* Determine different subsets of patients who benefit from these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to FAB subtype (refractory anemia (RA) or RA with ringed sideroblasts (RARS) vs RA with excess blasts (RAEB) vs RAEB in transformation (RAEB-t) vs juvenile myelomonocytic leukemia (JMML)).

Patients undergo complete medical and physical examination. Patients are screened for the following aberrations: -7, +8, +21, t(8;21), t(15;17), and inv(16). Smears of peripheral blood and bone marrow, as well as bone marrow biopsies and all cytogenetic and molecular studies performed on blood or bone marrow, are evaluated by a panel of international experts.

Patients with progressive RA or RARS undergo allogeneic stem cell transplantation (ASCT) according to EWOG-MDS SCT studies. Patients with stable RA or RARS wait for an optimal donor before undergoing ASCT. Patients with RAEB with fewer than 15% bone marrow blasts undergo ASCT. Patients with RAEB with at least 15% bone marrow blasts and patients with RAEB-t with fewer than 30% bone marrow blasts receive standard acute myeloid leukemia (AML) induction therapy and then undergo ASCT. Patients with RAEB-t with at least 30% bone marrow blasts are considered for standard AML induction therapy.

Patients with advanced JMML undergo evaluation for splenectomy and receive chemotherapy with mercaptopurine and cytarabine every 3-4 weeks (for 1-4 doses). Patients then undergo ASCT.

Patients are followed every 6 months.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically confirmed primary myelodysplastic syndromes (MDS)

  * Diagnosed between July 1, 1998 and June 30, 2002
* No prior aplastic anemia
* No prior congenital bone marrow failure syndrome, such as:

  * Fanconi's anemia
  * Kostmann syndrome
  * Shwachman syndrome
  * Dyskeratosis congenital
  * Amegakaryocytic thrombocytopenia
  * Diamond-Blackfan anemia
* No Down syndrome
* None of the following cytogenetic or molecular abnormalities:

  * t(8;21)(q22;q22)
  * t(15;17)(q22;q12)
  * inv(16)(p13;q22)
* No typical clinical and cytogenetic features of acute myeloid leukemia FAB M7 (i.e., acute megakaryocytic leukemia) with fewer than 30% blasts in bone marrow or peripheral blood

PATIENT CHARACTERISTICS:

Age

* Under 19

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Not specified

Renal

* Not specified

Other

* No other concurrent illness that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for MDS

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for MDS

Surgery

* Not specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1998-07

PRIMARY OUTCOMES:
Patient numbers in the different FAB subtypes

SECONDARY OUTCOMES:
Survival
Event-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Niemeyer, MD, Study Chair — Universitaetskinderklinik - Universitaetsklinikum Freiburg
Locations (1):
- Universitaetskinderklinik - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Germany

REFERENCES:
- [Derived] Drexler B, Schwarz-Furlan S, Baumann I, Rudelius M, Nollke P, Lebrecht D, Ramamoorthy S, Rotari N, Karow A, Hirabayashi S, Beier F, Behrens YL, Gohring G, Kalb R, Wlodarski MW, Strahm B, Erlacher M, Niemeyer CM, Yoshimi A. Long-term outcomes of patients with refractory cytopenia of childhood under observation only. Blood Adv. 2025 Aug 26;9(16):4279-4285. doi: 10.1182/bloodadvances.2025016136. PMID 40554414
- [Derived] Pastor VB, Sahoo SS, Boklan J, Schwabe GC, Saribeyoglu E, Strahm B, Lebrecht D, Voss M, Bryceson YT, Erlacher M, Ehninger G, Niewisch M, Schlegelberger B, Baumann I, Achermann JC, Shimamura A, Hochrein J, Tedgard U, Nilsson L, Hasle H, Boerries M, Busch H, Niemeyer CM, Wlodarski MW. Constitutional SAMD9L mutations cause familial myelodysplastic syndrome and transient monosomy 7. Haematologica. 2018 Mar;103(3):427-437. doi: 10.3324/haematol.2017.180778. Epub 2017 Dec 7. PMID 29217778
- [Derived] Gohring G, Michalova K, Beverloo HB, Betts D, Harbott J, Haas OA, Kerndrup G, Sainati L, Bergstraesser E, Hasle H, Stary J, Trebo M, van den Heuvel-Eibrink MM, Zecca M, van Wering ER, Fischer A, Noellke P, Strahm B, Locatelli F, Niemeyer CM, Schlegelberger B. Complex karyotype newly defined: the strongest prognostic factor in advanced childhood myelodysplastic syndrome. Blood. 2010 Nov 11;116(19):3766-9. doi: 10.1182/blood-2010-04-280313. Epub 2010 Aug 27. PMID 20802024